CLINICAL TRIAL: NCT02149784
Title: Palliative Resection of Asymptomatic Primary Tumor Following Effective Induction Chemotherapy in Colorectal Cancer Patients With Unresectable Distant Metastasis: a Multi-center, Prospective, Randomized Controlled Study
Brief Title: Effectiveness Study of Resection of Primary Tumor in Stage IV Colorectal Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gong Chen, Sun Yat-Sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140413
Record Dates: First submitted 2014-05-18; First posted 2014-05-29 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Metastasis colorectal cancer; Chemotherapy; Resection of primary tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical treatment group (Experimental): Unresectable mCRC patients who respond to chemotherapy will receive surgical resection of primary tumor.
  Interventions: Procedure: Surgical resection of primary tumor
- Chemotherapy group (No Intervention): Unresectable mCRC patients who were respond to chemotherapy will continue with chemotherapy.

INTERVENTIONS:
Procedure: Surgical resection of primary tumor — Surgical resection of primary tumor of mCRC patients who were respond to first line chemotherapy'
  Arms: Surgical treatment group

SUMMARY:
There is still no perfect treatment suggestion for patients with asymptomatic colorectal cancer with unresectable metastatic disease. Whether patients can benefit from palliative resection of primary tumor or not is still waiting for answer. The investigators hypothesis that asymptomatic metastatic colorectal cancer patients who respond to chemotherapy will benefit from primary tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* both genders
* ECOG:0-2 score
* Pathological confirmed colon cancer or rectal cancer with at least 12 cm far away from anal verge
* CT,MRI,or PET-CT confirmed metastasis
* MDT confirmed unresectable metastasis lesion
* No evidence of obstruction, bleeding, perforation
* WBC≥4.0×109/L，Neu ≥2.0×109/L，PLT≥100×109/L
* No contraindication for chemotherapy
* No evidence of other malignant tumor
* Expected survival time > 6 months

Exclusion Criteria:

* mCRC patients who did not respond to first line chemotherapy
* Require surgical intervention during the primary tumor-related symptoms
* Obvious coagulopathy
* Severe heart, liver, kidney damage or other serious uncontrolled medical illness or acute infection, cachexia
* Severe organ damage after chemotherapy, surgery or unable to continue to systemic chemotherapy
* Pregnant or lactating women or women of childbearing age who refuse to accept contraception.
* Nearly three months participated in clinical trials of other persons.
* Mental abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Number of Participants with Adverse Events both in surgery group and chemotherapy group | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gong Chen, Prof., Principal Investigator — Sun Yat-sen University; Zhi-zhong Pan, Prof., Study Chair — Sun Yat-sen University; De-Sen Wan, Prof., Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China